CLINICAL TRIAL: NCT00372216
Title: CIPAMI-Study: Clopidogrel Administered Prehospital to Improve Primary PCI in Patients With Acute Myocardial Infarction
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Stiftung Institut fuer Herzinfarktforschung (Other)
Collaborators: Bristol-Myers Squibb (Industry); Sanofi (Industry)
Responsible Party: Prof. Dr. Jochen Senges, Stiftung Institut fuer Herzinfarktforschung Ludwigshafen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CIPAMI
Record Dates: First submitted 2006-09-04; First posted 2006-09-06 (Estimated); Last update posted 2010-11-19 (Estimated); Status verified 2010-11

CONDITIONS: Myocardial Infarction
Keywords: myocardial infarction; Clopidogrel; primary PCI; TIMI-flow; STEMI within 6 hrs.
MeSH Terms: conditions — Myocardial Infarction | interventions — Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Pre-hospital loading dose of 600 mg Clopidogrel as early as possible (in addition to standard infarction therapy)
  Interventions: Drug: Clopidogrel (Iscover/Plavix)
- 2 (No Intervention): Standard infarction therapy (without study-specific additions, no Clopidogrel before angiography)

INTERVENTIONS:
Drug: Clopidogrel (Iscover/Plavix) — Pre-hospital loading-dose of 600 mg Clopidogrel as early as possible
  Other Names: Iscover 75 mg filmtablets; Plavix 75 mg filmtablets
  Arms: 1

SUMMARY:
Acute myocardial infarction is generally caused by a thrombotic occlusion of coronary arteries. Primary aim of early therapy is a fast and complete reperfusion of the infarcted myocardium, which can be achieved by either thrombolytic therapy or primary PCI.

Primary PCI is facilitated if the flow in the target vessel is restored prior to the intervention. In addition the results of recent trials hint that clinical outcome is improved by a patent infarct-vessel before primary PCI. The CIPAMI-study analyses the effect of an early administration of Clopidogrel on the flow-rates in subjects who suffered an acute myocardial infarction. For this purpose they are divided into two groups, both receiving standard baseline treatment. The subjects of one group additionally receive 600mg of Clopidogrel, as early as possible, while the subjects in the second group receive standard therapy. In the second group Clopidogrel is not allowed before initial angiography.

In both groups the flow-rates before and after PCI are analysed and compared in order to evaluate the efficacy, feasibility, and safety of the administration of a high loading dose Clopidogrel in the very early phase of STEMI in the prehospital setting.

ELIGIBILITY:
Inclusion Criteria:

* Acute STEMI <= 6 hrs.
* Planned percutaneous coronary intervention
* Age >= 18 years
* Ability to understand the natures, scope, and possible consequences of the study / legal capacity
* Informed consent

Exclusion Criteria:

* Thrombolytic therapy within 24 hours before randomization
* Effective oral or intravenous anticoagulation (INR>2, or PTT>2xcontrol)
* Known hemorrhagic diathesis
* Stroke or TIA within 3 months
* Evidence of an active gastrointestinal or urogenital bleeding
* Major surgery (including CABG) within 6 weeks
* Contraindication to Clopidogrel
* Severe renal or hepatic insufficiency
* Contraindication to coronary angiography
* Planned administration of a GP IIb/IIIa-Inhibitor before angiography
* Pregnant or nursing (lactating) women
* Women with childbearing potential
* Patients currently (within the last 10 days) treated with clopidogrel or ticlopidine
* Participation in another clinical or device trial within the previous 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 337 (Actual)
Dates: Start 2006-10; Primary Completion 2009-10 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
TIMI 2/3 patency of the infarct-related artery immediately prior to PCI | Assessment at primary PCI, asap after inclusion of the subject

SECONDARY OUTCOMES:
TIMI 3 patency before PCI | Assessment before primary PCI, asap after inclusion of the subject
TIMI 3 patency after PCI | Assessment at primary PCI, asap after inclusion of the subject
ST resolution immediately before angiography and 60-90 minutes after PCI | Assessment immediately before angiography until 90 minutes after PCI
Death, re-MI, urgent revascularisation until 48 hours and until hospital discharge | Starting with inclusion of the subject until day 7
Stroke (hemorrhagic, non-hemorrhagic) | Starting with inclusion of the subject until day 7
Severe bleeding complications according to the TIMI classification | Starting with inclusion of the subject until day 7

CONTACTS AND LOCATIONS:
Overall Officials: Uwe Zeymer, MD, Principal Investigator — Klinikum der Stadt Ludwigshafen, Med. Klinik B, Ludwigshafen Germany
Locations (25):
- Austria (3):
  - Universitaetsklinikum Innsbruck, Innsbruck
  - Hanusch-Krankenhaus, Vienna
  - Wilhelminenspital, Vienna
- Germany (22):
  - Universitaetsklinikum Mannheim, Mannheim, Baden-Wurttemberg
  - Staedtisches Klinikum, Brandenburg, Brandenburg
  - KMG-Kliniken AG / Klinikum Wittstock, Wittstock, Brandenburg
  - Kerckhoff Klinik, Bad Nauheim, Hesse
  - Klinikum Darmstadt, Darmstadt, Hesse
  - Klinikum der Johann-Wolfgang-Goethe Universitaet, Frankfurt am Main, Hesse
  - Universitaetsklinikum Giessen, Giessen, Hesse
  - Kreiskrankenhaus Bergstrasse, Heppenheim an der Bergstrasse, Hesse
  - St. Vincenz-Krankenhaus, Limburg an der Lahn, Hesse
  - Allgemeines Krankenhaus, Celle, Lower Saxony
  - Evangelisches Krankenhaus, Holzminden, Lower Saxony
  - Städtisches Klinikum, Lüneburg, Lower Saxony
  - Universitaetsklinikum Rostock, Rostock, Mecklenburg-Vorpommern
  - Klinikum Leverkusen, Leverkusen, North Rhine-Westphalia
  - Klinikum der Stadt Ludwigshafen, Med. Klinik B, Ludwigshafen am Rhein, Rhineland-Palatinate
  - Klinikum Saarbruecken, Saarbrücken, Saarland
  - Universitaet Leipzig - Herzzentrum, Leipzig, Saxony
  - Sana Klinikum Lichtenberg / Oskar-Ziethen-Krankenhaus, Berlin, State of Berlin
  - Universitaetsklinikum Benjamin Franklin, Berlin, State of Berlin
  - Vivantes Klinikum Neukoelln, Berlin, State of Berlin
  - Maria Heimsuchung / Caritas-Klinik Pankow, Berlin, State of Berlin
  - DRK-Kliniken Westend, Berlin, State of Berlin